CLINICAL TRIAL: NCT06638112
Title: Comparison of Postoperative Quality of Recovery by Anesthetic Method in Patients Undergoing Shoulder Arthroscopy: Brachial Plexus Block for Pain Control Under General Anesthesia Versus Brachial Plexus Block for Surgical Block Under Sedation
Brief Title: Comparison of Postoperative Quality of Recovery by Anesthetic Method in Patients Undergoing Shoulder Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2408-076-1562
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Shoulder Arthroscopy
MeSH Terms: interventions — Brachial Plexus Block; Anesthesia, General; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel group, open-label randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General anesthesia (Active Comparator): The patient undergoes shoulder arthroscopy under general anesthesia after receiving a preoperative brachial plexus block for intra- and postoperative analgesia.
  Interventions: Procedure: General Anesthesia (control group)
- Brachial plexus block (Experimental): The patient undergoes shoulder arthroscopy under brachial plexus block and intraoperative sedation with remimazolam or propofol.
  Interventions: Procedure: Brachial Plexus Block

INTERVENTIONS:
Procedure: Brachial Plexus Block — Interscalene brachial plexus block with 0.75% ropivacaine. Intraoperative sedation with remimazolam or propofol.
  Arms: Brachial plexus block
Procedure: General Anesthesia (control group) — General anesthesia with propofol, fentanyl and rocuronium for induction, and with sevoflurane for maintenance. Brachial plexus block with 0.5% ropivacaine for intra- and postoperative analgesia.
  Arms: General anesthesia

SUMMARY:
The aim of this study is to compare the quality of recovery in patients undergoing arthroscopic shoulder surgery depending on the type of anesthesia used:

1. general anesthesia with preoperative brachial plexus block for intra- and postoperative analgesia
2. regional anesthesia (brachial plexus block) with intraoperative sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 19 years and above, scheduled for shoulder arthroscopic surgery

Exclusion Criteria:

* emergency operation
* inflammation or infection at the site of nerve block administration
* inability to perform the quality of recovery questionnaire due to dementia or delirium
* severe lung disease (e.g. chronic obstructive pulmonary disease or interstitial lung disease)
* contraindication to brachial plexus block
* history of hypersensitivity or side effect to ropivacaine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery (QoR-15) at 48 hours post-surgery | at 48 hours post-surgery
  Quality of recovery (QoR-15) at 48 hours post-surgery (0-150)

SECONDARY OUTCOMES:
Antiemetic administration | rom end of surgery up to 48 hours post-surgery
  Antiemetic administration from end of surgery up to 48 hours post-surgery
Baseline hemidiagphramatic paralysis | On the day of surgery, before the operation
  Baseline hemidiagphramatic paralysis
Postoperative hemidiagphramatic paralysis | Immediately after surgery
  Postoperative hemidiagphramatic paralysis
Quality of recovery (QoR-15) on the day before surgery | on the day before surgery
  Quality of recovery (QoR-15) on the day before surgery (0-150)
Quality of recovery (QoR-15) 24 hours post-surgery | at 24 hours post-surgery
  Quality of recovery (QoR-15) 24 hours post-surgery (0-150)
Postoperative pain 1 hour post-surgery | at 1 hour post-surgery
  Postoperative pain 1 hour post-surgery (Numeric rating scale, 0: no pain; 10: worst pain imaginable)
Postoperative pain 6 hours post-surgery | at 6 hours post-surgery
  Postoperative pain 6 hours post-surgery (Numeric rating scale, 0: no pain; 10: worst pain imaginable)
Postoperative pain 12 hours post-surgery | at 12 hours post-surgery
  Postoperative pain 12 hours post-surgery (Numeric rating scale, 0: no pain; 10: worst pain imaginable)
Postoperative pain 24 hours post-surgery | at 24 hours post-surgery
  Postoperative pain 24 hours post-surgery (Numeric rating scale, 0: no pain; 10: worst pain imaginable)
Postoperative pain 48 hours post-surgery | at 48 hours post-surgery
  Postoperative pain 48 hours post-surgery (Numeric rating scale, 0: no pain; 10: worst pain imaginable)
Incidence of postoperative nausea and/or vomiting (PONV) 1 hour post-surgery | at 1 hour post-surgery
  Incidence of postoperative nausea and/or vomiting (PONV) 1 hour post-surgery
Incidence of postoperative nausea and/or vomiting (PONV) 6 hours post-surgery | at 6 hours post-surgery
  Incidence of postoperative nausea and/or vomiting (PONV) 6 hours post-surgery
Incidence of postoperative nausea and/or vomiting (PONV) 12 hours post-surgery | at 12 hours post-surgery
  Incidence of postoperative nausea and/or vomiting (PONV) 12 hours post-surgery
Incidence of postoperative nausea and/or vomiting (PONV) 24 hours post-surgery | at 24 hours post-surgery
  Incidence of postoperative nausea and/or vomiting (PONV) 24 hours post-surgery
Incidence of postoperative nausea and/or vomiting (PONV) 48 hours post-surgery | at 48 hours post-surgery
  Incidence of postoperative nausea and/or vomiting (PONV) 48 hours post-surgery
Rescue opioid analgesic administration | from end of surgery up to 48 hours post-surgery
  Rescue opioid analgesic administration from end of surgery up to 48 hours post-surgery (morphine milligram equivalent, MME)

CONTACTS AND LOCATIONS:
Overall Officials: Hansol Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided